CLINICAL TRIAL: NCT06175455
Title: Diaphragm Dysfunction After COVID-19 as Determined by Dynamic Chest Radiography
Acronym: DD-COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-537
Record Dates: First submitted 2023-12-14; First posted 2023-12-19 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Long Covid19
Keywords: coronavirus; diaphragm dysfunction; dynamic chest radiography; dyspnea
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Coronavirus Infections; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: Healthy, age and sex matched controls
  Interventions: Device: dynamic chest radiography
- Long Covid: patients who experienced persistent respiratory symptoms four weeks after contracting COVID-19
  Interventions: Device: dynamic chest radiography

INTERVENTIONS:
Device: dynamic chest radiography — A recent technological advancement in this field is dynamic chest radiography (DCR), which is a low-dose imaging system capable of producing continuous moving images

SUMMARY:
Dynamic chest radiography (DCR) is a rapid and easily performed technique that captures real-time continuous images of the moving chest. COVID-19 has led to various complications and long-term effects, with dyspnea being a common symptom experienced by many patients. Studies conducted abroad have indicated that dyspnea following a new coronavirus infection can be attributed to diaphragm dysfunction. This study using DCR aims to describe diaphragm function in patients after coronavirus disease (COVID-19).

DETAILED DESCRIPTION:
It has been estimated that approximately 80% of individuals infected with the new coronavirus will experience one or more long-term symptoms following recovery, with dyspnea being a frequent clinical complaint. However, this dyspnea cannot be adequately made clear by conventional clinical diagnostic measures, including pulmonary function tests and cardiac evaluation.

Currently, 9 clinical studies have explored the relationship between diaphragm dysfunction and COVID-19 in a small number of samples. To evaluate diaphragmatic function, there are several examination methods currently available including transdiaphragmatic pressure measurement, diaphragmatic ultrasound, and neuroelectrophysiological examination. However, these methods pose challenges in terms of implementation and widespread use, as they require a considerable amount of time and user experience. Therefore, there is a substantial unmet clinical demand for these methods.

A recent technological advancement in this field is dynamic chest radiography (DCR), which is a low-dose imaging system capable of producing continuous moving images. Compared to traditional fluoroscopic techniques, dynamic chest radiography offers several advantages, including simplicity of operation, reduced radiation dose, and the ability to provide quantitative data on diaphragm and chest wall motion. It has been used to diagnose diaphragmatic dysfunction by effectively identifying paradoxical diaphragmatic movement.

In this study, patients who experienced persistent respiratory symptoms four weeks after COVID-19 underwent DCR to observe diaphragm function and determine its relationship to dyspnea and clinical detection. This research marks the first instance of using DCR to investigate diaphragm dysfunction following COVID-19. The study shows promising research potential in understanding the role of diaphragm abnormalities and addressing the limitations of traditional examination methods for assessing diaphragm function.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 group:

  1. Voluntarily sign the informed consent form;
  2. Aged equal to or older than 18 years old, regardless of gender;
  3. Inpatients with COVID-19 who mainly complain of dyspnea, dyspnea If it persists or develops and lasts for more than 4 weeks after acute COVID-19, it is related to long COVID-19; (confirmed infection with COVID-19 through nucleic acid monitoring or hospital laboratory data);
  4. Lung function measurements have been completed during hospitalization due to diagnosis and treatment needs;
  5. Be able to cooperate in completing the dynamic chest X-ray (complete the positioning of the dynamic chest X-ray for 20 seconds, and breathe calmly and forcefully during this period; be able to hold breath for at least 7 seconds).
* Control group:

  1. Voluntarily sign the informed consent form;
  2. Aged equal to or older than 18 years old, regardless of gender;
  3. People from the health examination center, and the age, gender are matched in the COVID-19 group and have no previous acute or chronic cardiopulmonary disease, no abnormalities in previous lung physical examinations and lung imaging examinations, and no history of infectious diseases in the past month;
  4. Physical examination items are required People who are suitable for ordinary chest X-ray examination;
  5. Be able to cooperate in completing dynamic chest X-ray (complete dynamic chest X-ray positioning for 20 seconds, during which period, breathe calmly and forcefully, and be able to hold breath for at least 7 seconds).

Exclusion Criteria:

* COVID-19 group:

  1. Not suitable to participate in this study;
  2. Combined with serious life-threatening diseases, such as cardiovascular and cerebrovascular diseases, lung cancer, airway obstruction, etc.;
  3. Combined with pneumothorax, pulmonary insufficiency, chronic disease, interstitial disease, lung surgery history or recent planned surgery;
  4. Mental disorder and unable to cooperate with the operator;
  5. Pregnant or lactating women;
  6. Major radiation related to the research within 12 months before consent Exposure (participating in previous studies involving radiation exposure, the research dose is limited to 0.4mSv);
  7. No evidence of having been infected with the new coronavirus;
  8. Unable to cooperate in completing dynamic chest X-rays;
  9. Unable to complete lung function measurements；
* Control group:

  1. Not suitable to participate in this study;
  2. Patients with previous acute or chronic cardiopulmonary disease, previous lung physical examination, lung imaging examination abnormalities, within the past 1 month Have a history of infectious diseases;
  3. Mentally abnormal and unable to cooperate with the operator;
  4. Pregnant or lactating women;
  5. Significant radiation exposure related to the research within 12 months before consent (participation in previous research involving radiation exposure, The study dose is limited to 0.4mSv); 6) Unable to cooperate in completing dynamic chest X-ray;.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will compare a group of adults (over 18 years) in the community who experience breathlessness as a result of long COVID with a control group of healthy volunteers who are matched in terms of age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
diaphragm assessment | 5 months
  observe the differences in dynamic chest X-ray measurements between patients with COVID-19 and normal people

SECONDARY OUTCOMES:
Correlation between lung function and DCR | 5 months
  observe the correlationbetween lung function and DCR

CONTACTS AND LOCATIONS:
Overall Officials: Liu Laiyu, professor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Yudong, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No